## Mayo Clinic: Office for Human Research Protection Oral Consent Script

Protocol Title: Dual-plane ultrasound imaging during vascular access procedures.

IRB #: 19-008071

Principal Investigator: Robert Anderson DNP, ARNP, CNP

You are being asked to participate in a research study which will evaluate the use of a dual-view ultrasound probe to assist in placement of the arterial line that will be used to monitor your blood pressure during surgery. An arterial line would be placed as standard care.

If you agree to participate a member of the anesthesia team will use a ultrasound probe which provides them two different views of the artery to help guide the arterial catheter into the artery. Ultrasound is used to place arterial catheters; however typical ultrasound probes provide the operator with only one view. This ultrasound probe allows the operator to see the artery in two dimensions to assist them in placing the arterial catheter.

A standard arterial catheter and procedure of placement will be utilized; the only modification to the procedure is the use of a dual-view as compared to a single-view ultrasound probe.

If you decide to participate, you will need to read and sign the Authorization to Use and Disclose Protected Health Information (HIPAA) form and return it with the questionnaire. We are not allowed to use the answers without your signature on the HIPAA form. An extra copy is included for your records.

The risks of this research study are minimal, which means that we do not believe that they will be any different than what you would experience at a routine clinical visit or during your daily life. You may refuse to answer any survey question(s) that you do not wish to answer.

This study will not make your health better but has the potential to improve efficiency and success rates of arterial catheter placement. It is for the benefit of research.

Your information collected as a part of this research, will not be used or distributed for future research studies, even if identifiers are removed.

Please understand your participation is voluntary and you have the right to withdraw your consent or discontinue participation at any time without penalty. Specifically, your current or future medical care at the Mayo Clinic will not be jeopardized if you choose not to participate.

If you have any questions about this research study you can contact me at 507-266-7513. If you have any concerns, complaints, or general questions about research or your rights as a participant, please contact the Mayo Institutional Review Board (IRB) to speak to someone independent of the research team at 507-266-4000 or toll free at 866-273-4681.

 $https://mctools-my.sharepoint.com/personal/anderson\_robert2\_mayo\_edu/Documents/H\_Mig/Dual-view\ US\ Probe/21-007039\ Oral\ consent\ for\ patients\ 07122021.doc \\ Page\ 1\ of\ 1$ 

Master copies are retained online. Printed copies are considered current only on the date printed, unless stamped ORIGINAL or COPY in red ink.